CLINICAL TRIAL: NCT01469481
Title: An Open Label, Single-Period, Phase 1 Study To Evaluate The Pharmacokinetics, Excretion, Mass Balance And Metabolism Of [14c]-PF-04991532 In Healthy Adult Male Subjects
Brief Title: Single Dose Study To Study The Absorption, Metabolism And Excretion Of PF-04991532
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B2611007
Record Dates: First submitted 2011-10-28; First posted 2011-11-10 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: diabetes mellitus; ADME
MeSH Terms: conditions — Diabetes Mellitus | interventions — 6-(3-cyclopentyl-2-(4-(trifluoromethyl)-1H-imidazol-1-yl)propanamido)nicotinic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-04991532

INTERVENTIONS:
Drug: PF-04991532 — a single oral dose of [14C]PF-04991532 (450 mg/100 uCi suspension)

SUMMARY:
The purpose of this study is to evaluate the excretion balance, metabolic profile and the routes of excretion of [14C]PF-04991532 in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg(110 lbs).
* An informed consent document signed and dated by the subject.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or clinical findings at Screening.
* History of irregular bowel movements (eg, irritable bowel syndrome or frequent episodes of diarrhea or constipation).
* Any condition possibly affecting drug absorption (eg, appendectomy, gastrectomy).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Mass Balance: Urinary and fecal excretion of radioactivity over time expressed as a percentage of the total radioactive dose administered. | 0-168 hrs
Metabolic Profiling/identification and determination of relative abundance of PF-04991532 and the metabolites of PF-04991532 in plasma, urine, and feces. | 0-168 hrs
radioactivity AUC | 0-168 hrs
plasma PF-04991532 AUC | 0-168 hrs
radioactivity Cmax | 0-168 hrs
plasma PF-04991532 Cmax | 0-168 hrs
plasma PF-04991532 Tmax | 0-168 hrs
radioactivity Tmax | 0-168 hrs
plasma PF-04991532 t1/2 | 0-168 hrs
radioactivity t1/2 | 0-168 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Tacoma, Washington, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2611007&StudyName=Single%20Dose%20Study%20To%20Study%20The%20Absorption%2C%20Metabolism%20And%20Excretion%20Of%20PF-04991532